CLINICAL TRIAL: NCT04898972
Title: Mindfulness-based Stress Reduction Intervention in Patients With COPD and Their Caregivers
Brief Title: Mindfulness-based Intervention in COPD Dyads
Acronym: MIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Maria Matarese, Associate Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29.17 OSS ComEt CBM
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyad; caregiver; mindfulness; COPD; patient; intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction intervention (Experimental): Patient-family caregiver dyads will take part in 8-week Mindfulness-based stress reduction intervention (MBSR).
  Interventions: Behavioral: Mindfulness-based stress reduction intervention
- information booklet (Active Comparator): Patient-informal caregiver dyads will receive an informative booklet on stress reduction strategies
  Interventions: Behavioral: Information on stress reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction intervention — The 8-group sessions of MBSR will be conducted once a week, lasting two and a half hours, with two additional sessions in the following two months. Between sessions, participants will have to practice at home for 45 minutes a day, 6 days a week. For the practice, patients and caregivers will be provided with audio files containing the meditations proposed in the classroom, readings, and the diary of the practice. During the sessions, the following mindfulness-based techniques will be introduced: body scan; sitting meditation; awareness movement exercises; and walking meditation.The sessions will be held face to face or online using common videoconferencing platforms, such as Skype or Zoom, based on the preferences of the participants. This will facilitate the participation of patients and caregivers, overcoming the obstacles related to travel. The course will be taught by certified mindfulness teachers with experience in MBSR interventions on patients with respiratory diseases.
  Arms: Mindfulness-based stress reduction intervention
Behavioral: Information on stress reduction — COPD patient-caregiver dyads will be delivered by hand, sent by email or by post an information booklet "Coping with your chronic disease", targeting COPD patients, to teach them how to manage stress. This booklet, available in Italian, provides simple information on the meaning of stress and anxiety, and suggests some actions that people can implement at home to reduce stress.
  Arms: information booklet

SUMMARY:
This study evaluates the effectiveness of a Mindfulness-Based Stress Reduction intervention (MBSRI) on the reduction of stress, anxiety, and depression in people with COPD and their family caregivers. The experimental group will receive the MBSRI and the control group an informational intervention on stress management.

DETAILED DESCRIPTION:
People affected by Chronic Obstructive Pulmonary Disease (COPD) and their family caregivers (named dyads) often suffer from psychological distress, because of the physical problems and social isolation imposed by the disease. Such psychological distress can influence the ability of patients and caregivers to manage the disease. Mindfulness-based interventions have showed benefits in improving the psychological status in various clinical situations. A 8-week mindfulness based-stress reduction intervention will be offered to a group of COPD patient-caregiver dyads and its effectiveness will be assessed comparing the effects on a control group to whom an informational intervention on stress reduction will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Persons able to read and understand Italian.
* people affected by COPD stage C (GOLD 3 o 4, and/or 2 or more exacerbations per year or 1 or more hospitalizations for exacerbations and score of COPD assessment test-CAT < 10 or mMRC 0-1).
* People affected by COPD stage D (GOLD 3 o 4, and/or 2 or more exacerbations per year or 1 or more hospitalizations for exacerbations and score of COPD assessment test-CAT ≥ 10 or mMRC ≥ 2).

Exclusion Criteria:

* Persons or dyads not able to guarantee the presence on the MBSR intervention sessions for the four months requested.
* Persons with diagnosis of anxiety or depression.
* Persons that have practiced before or actually practice yoga or mindfulness.
* Persons with cognitive impairment.
* Persons under continuous oxygen therapy.
* Persons with diagnosis of cancer or other terminal diseases or any psychiatric problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in perceived stress measured by Perceived Stress Scale (PSS) at 8 weeks and 16 weeks | at baseline, after 8 weeks, and after 16 weeks from baseline
  The perceived stress entails the feelings or thoughts that an individual has about how much stress they are under at a given point in time. It will be measured in patients and caregivers using the Perceived Stress Scale (PSS) that is a 10 item-self-report instrument: its score ranges from 0 to to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Change = (8 weeks- baseline scores) (16 weeks-baseline scores), and (16-weeks-8 weeks scores).
Change from baseline in anxiety level measured by Generalized Anxiety Disorder scale (GAD-7) at 8 weeks and 16 weeks. | at baseline, after 8 weeks, and after 16 weeks from baseline
  The anxiety level will be measured in patients and caregivers using the 7-item Generalized Anxiety Disorder scale (GAD-7). Its scores range from 0 to 21. Cut points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety. Change = (8 weeks- baseline scores) (16 weeks-baseline scores), and (16-weeks-8 weeks scores).
Change from baseline in depression measured by Patient Health Questionnaire (PHQ-9) at 8 weeks and 16 weeks | at baseline, after 8 weeks, and after 16 weeks from baseline
  The depressive symptoms in patients and caregivers will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Its score range from 0 (no symptoms) to 27 (nearly daily symptoms). Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. Change = (8 weeks- baseline scores) (16 weeks-baseline scores), and (16-weeks-8 weeks scores).

SECONDARY OUTCOMES:
Change from baseline in subjective quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI) at 8 and 16 weeks. | at baseline, after 8 weeks, and after 16 weeks from baseline
  The quality and patterns of sleep in patients and caregivers will be measured by PSQI that is a self-report questionnaire measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. The global score ranges from 0 to 21, the higher the score, the worse the sleep quality. A global score of 5 or more indicates poor sleep quality; Change = (8 weeks- baseline scores) (16 weeks-baseline scores), and (16-weeks-8 weeks scores).
Change from baseline in mindfulness experience measured by Five Facet Mindfulness Questionnaire (FFMQ) at 8 and 16 weeks. | at baseline, after 8 weeks, and after 16 weeks from baseline
  The mindfulness abilities in patients and caregivers will be measured by a self-reported questionnaire, FFMQ, that comprises 39 items assessing five facets of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Higher global score shows a higher mindfulness disposition. Change = (8 weeks- baseline score), (16 weeks-baseline scores), and (16 weeks-8 weeks scores).
Change in health-related quality of life measured by Short Form 12 Health Survey (SF-12) at 8 and 16 weeks | at baseline, after 8 weeks, and after 16 weeks from baseline
  The physical and mental health-related quality of life of patients and caregivers will by measured by the SF-12 that comprises 12 items. Higher the scores the better the quality of life. Change = (8 weeks- baseline scores), (16 weeks-baseline scores), and (16 weeks-8 weeks scores).
Change in impact of the COPD on patient's life measured by COPD Assessment Test (CAT) at 8 weeks and 16 weeks | at baseline, after 8 weeks, and after 16 weeks from baseline
  The CAT is a 8-item instrument that assesses health-related quality of life and symptom burden in COPD patients. Range of CAT scores from 0-40. Higher scores denote a more severe impact. Change = (8 weeks- baseline scores), (16 weeks-baseline scores), and (16 weeks-8 weeks scores).
Change in patient's dyspnea measured by the Modified Medical Research Council scale (mMRC) at 8 and 16 weeks | at baseline, after 8 weeks, and after 16 weeks from baseline
  The mMRC is a 5-point (0-4) scale that will be used to measure the severity of dyspnea in patients. Higher scores mean worse dyspnea. Change = (8 weeks-baseline scores), (16 weeks-baseline scores), and (16 weeks-8 weeks scores).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Matarese, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Campus Bio-medico University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that will be used in the result publications.
Supporting Information: SAP, ICF
Time Frame: From the date of study publication up to 4 years later
Access Criteria: Formal request by email from researchers affiliated to university centers

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chan RR, Giardino N, Larson JL. A pilot study: mindfulness meditation intervention in COPD. Int J Chron Obstruct Pulmon Dis. 2015 Mar 2;10:445-54. doi: 10.2147/COPD.S73864. eCollection 2015. PMID 25767382
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Harrison SL, Lee A, Goldstein RS, Brooks D. Perspectives of healthcare professionals and patients on the application of mindfulness in individuals with chronic obstructive pulmonary disease. Patient Educ Couns. 2017 Feb;100(2):337-342. doi: 10.1016/j.pec.2016.08.018. Epub 2016 Aug 20. PMID 27567496
- [Background] Harrison SL, Lee A, Janaudis-Ferreira T, Goldstein RS, Brooks D. Mindfulness in people with a respiratory diagnosis: A systematic review. Patient Educ Couns. 2016 Mar;99(3):348-355. doi: 10.1016/j.pec.2015.10.013. Epub 2015 Oct 23. PMID 26561308
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Mularski RA, Munjas BA, Lorenz KA, Sun S, Robertson SJ, Schmelzer W, Kim AC, Shekelle PG. Randomized controlled trial of mindfulness-based therapy for dyspnea in chronic obstructive lung disease. J Altern Complement Med. 2009 Oct;15(10):1083-90. doi: 10.1089/acm.2009.0037. PMID 19848546
- [Background] Pbert L, Madison JM, Druker S, Olendzki N, Magner R, Reed G, Allison J, Carmody J. Effect of mindfulness training on asthma quality of life and lung function: a randomised controlled trial. Thorax. 2012 Sep;67(9):769-76. doi: 10.1136/thoraxjnl-2011-200253. Epub 2012 Apr 27. PMID 22544892
- [Background] Clari, M., Conti, A., Fontanella, R., Rossi, A., & Matarese, M. (2020). Mindfulness-based programs for people with chronic obstructive pulmonary disease: a mixed methods systematic review. Mindfulness, 1-20.